CLINICAL TRIAL: NCT04975256
Title: A Phase 1/1b Trial of MRTX849 in Combination With BI 1701963 in Patients With Advanced Solid Tumors With KRAS G12C Mutation
Brief Title: Adagrasib in Combination With BI 1701963 in Patients With Cancer (KRYSTAL 14)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision was made to terminate this study to further enrollment, as of 08 March 2022. The decision was made primarily due to a change in development strategy.
Sponsor: Mirati Therapeutics Inc. (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 849-014
Expanded Access: NCT05162443 (Approved for marketing)
Record Dates: First submitted 2021-07-06; First posted 2021-07-23 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Advanced Cancer; Metastatic Cancer; Malignant Neoplasm of Colon; Malignant Neoplasm of Lung; Malignant Neoplastic Disease
Keywords: KRAS G12C; SOS1 Inhibitor; NSCLC; CRC; Non Small Cell Lung Cancer; Colon Cancer; Advanced Solid Tumor; Metastatic Cancer; Pancreatic Cancer; adagrasib
MeSH Terms: conditions — Neoplasm Metastasis; Colonic Neoplasms; Lung Neoplasms; Neoplasms; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms | interventions — adagrasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Experimental): Dose escalation of MRTX849 and BI 1701963 to determine maximum tolerated dose in combination
  Interventions: Drug: MRTX849; Drug: BI 1701963
- Dose expansion (Experimental): Expansion cohorts in NSCLC and CRC patients to ensure sufficient safety experience, pharmacokinetic information, and early evidence of clinical activity of MRTX849 in combination with BI 1701963
  Interventions: Drug: MRTX849; Drug: BI 1701963

INTERVENTIONS:
Drug: MRTX849 — KRAS G12C inhibitor
  Other Names: KRAS G12C inhibitor; adagrasib
Drug: BI 1701963 — SOS1 Inhibitor
  Other Names: SOS1 Inhibitor

SUMMARY:
This study will evaluate safety, tolerability, drug levels, molecular effects and clinical activity of MRTX849 (adagrasib) in combination with BI 1701963 in patients with advanced solid tumors that have a KRAS G12C mutation.

DETAILED DESCRIPTION:
This study will evaluate safety, tolerability, pharmacokinetics, metabolites, pharmacodynamics and clinical activity of MRTX849 (adagrasib) in combination with BI 1701963 in patients with advanced solid tumors with a KRAS G12C mutation. MRTX849 is an orally available small molecule inhibitor of KRAS G12C and BI 1701963 is a SOS1 pan-KRAS inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a solid tumor malignancy with KRAS G12C mutation (phase 1b must be either Non-Small Cell Lung Cancer or Colorectal Cancer)
* Unresectable or metastatic disease
* No available treatment with curative intent
* Adequate organ function

Exclusion Criteria:

* History of intestinal disease, inflammatory bowel disease, major gastric surgery, or other gastrointestinal conditions likely to alter absorption of study treatment or result in inability to swallow
* Other active cancer
* Cardiac abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Characterize the number of patients with treatment emergent adverse events of the combination regimen in patients with advanced solid tumor malignancies with KRAS G12C mutation | 20 months
  Number of participants with treatment related adverse events
Evaluate Pharmacokinetics of the combination regimen | 20 months
  Blood plasma concentration
Establish Maximum Tolerated Dose | 12 months
  Number of patients with dose limiting toxicity

SECONDARY OUTCOMES:
Evaluate preliminary clinical activity of the combination regimen | 20 months
  Objective response rate in accordance with Response Evaluation Criteria in Solid Tumors (RECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Chao, MD, Study Director — Mirati Therapeutics
Locations (4):
- United States (4):
  - Washington University School of Medicine, St Louis, Missouri
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Next Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No